CLINICAL TRIAL: NCT02190851
Title: Evaluation of Treatment by Transcutaneous Electrical Nerve Stimulation (TENS) of the Posterior Tibial Nerve for Lower Urinary Tract Disorders in Parkinson's Syndrome
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Lower Urinary Tract Disorders in Parkinson's Syndrome
Acronym: UROPARKTENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13 7047 01; 13-0147 (Other Grant/Funding Number: French Ministry of Health, PHRC 2013)
Record Dates: First submitted 2014-07-08; First posted 2014-07-15 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2020-11

CONDITIONS: Parkinson's Disease
Keywords: urinary disorders; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- electrical nerve stimulation (TENS) (Experimental): Two electrodes are attached around the internal malleolus and connected to the TENS unit, by UROSTIM 2.
  The sessions last 20 minutes daily (frequency 10Hz, duration 200µs), at maximum intensity of painless stimulation, every day at the same time, on the right side for 3 months.
  Interventions: Device: TENS
- Control group (Placebo Comparator): The device will have been previously set to deliver a stimulation below the effective threshold. In all cases, the device displays 20mA. Stimulation sessions are 20 minutes daily, every day at the same time, on the right side for 3 months.
  Interventions: Device: Control

INTERVENTIONS:
Device: TENS — Two electrodes are attached around the internal malleolus and connected to the TENS unit.
  The sessions last 20 minutes daily (frequency 10Hz, duration 200µs), at maximum intensity of painless stimulation, every day at the same time, on the right side for 3 months.
  Other Names: UROSTIM 2 by SchwaMedica
  Arms: electrical nerve stimulation (TENS)
Device: Control — The device will have been previously set to deliver a stimulation below the effective threshold. In all cases, the device displays 20mA. Stimulation sessions are 20 minutes daily, every day at the same time, on the right side for 3 months.
  Arms: Control group

SUMMARY:
Only one study has evaluated the effect of TENS in LUTD in Parkinson's syndromes. It was reported at the congress of the "Société Interdisciplinaire Francophone d'UroDynamique et de Pelvi-Perinéologie" (SIFUD-PP) in 2011 by Ohanessian et al., and comprised 6 female patients with Parkinson's disease (PD) or multisystem atrophy (MSA), with overactive bladder. Transcutaneous electrical nerve stimulation, 20 minutes daily for 6 weeks, was associated with subjective improvement of LUTD assessed with the Patient Global Impression of Improvement (PGI-I) in 5 of the 6 patients.

In view of the encouraging results of this pilot study, we hypothesize that TENS treatment may improve LUTD in patients with a Parkinson's syndrome, Parkinson's disease (PD) and multisystem atrophy (MSA).

DETAILED DESCRIPTION:
The principal objective is to compare the efficacy of transcutaneous electrical nerve stimulation of the posterior tibial nerve with placebo stimulation, applied 20 minutes daily for 3 months, in Lower Urinary Tract Disorders (LUTD) in patients with Parkinson's disease or multisystem atrophy, evaluated using the PGI-I (Patient Global Impression of improvement) tool.

The secondary objectives are to compare the efficacy of TENS with placebo stimulation on change before/after 3 months of treatment on:

* the intensity of urinary symptoms, evaluated using the Patient Global Impression of Severity (PGI-S) scale
* the number of voidings in 24 hours, number of episodes of urinary incontinence in 24 hours and maximum bladder capacity, evaluated by a voiding diary over 3 days
* urinary symptoms, evaluated with the urinary symptom profile (USP) questionnaire
* quality of life, assessed by the Qualiveen-SF® questionnaire
* post-void residual volume measured by bladder ultrasound and effect on the development of infectious complications, by comparing the number of urinary infections over 3 months in each group.

Lastly, the safety of TENS will be compared with that of placebo stimulation by the occurrence of adverse events during the 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Parkinson disease or multisystem atrophy
* Refractory lower urinary tract disorders or contra-indications or intolerance to the usual oral treatments
* Patient capable of completing the questionnaires
* Patient whose written informed consent has been obtained
* Patient registered with a social security scheme

Exclusion Criteria:

* Pregnancy and breast-feeding
* Contra-indications to TENS (local skin problems, metal ankle joint replacement, cardiac pacemaker, peripheral neuropathy, subthalamic deep brain stimulation)
* Associated neurological disorders (stroke, dementia, multiple sclerosis, spinal cord lesions, peripheral neuropathy) or urological disorders (bladder outlet obstruction, cancer, pelvic organ prolapse, interstitial cystitis)
* Unilateral neurological disability
* Legally incompetent patient, patient under legal protection
* Participation in another study during the present study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Improvement Score Measure | 3 months
  The score is measured after 3 months treatment

SECONDARY OUTCOMES:
Patient global Impression of severity score measure | december 1, 2014
  the patient self-assesses the severity of his lower urinary tract disorders

CONTACTS AND LOCATIONS:
Overall Officials: Xavier GAME, MD, Principal Investigator — University Hospital, Toulouse
Locations (11):
- France (11):
  - Clinique Saint Augustin, Bordeaux
  - Hospital Chenevier, Créteil
  - Hospital Poincare, Garches
  - Huriez Hospital, Lille
  - University Hospital, Lyon
  - Uiversity hospital, Marseille
  - University hospital, Paris
  - Hospital Dubos, Pontoise
  - Pontchaillou Hospital, Rennes
  - University hospital, Rouen
  - UHToulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Castel-Lacanal E, Game X, Clanet M, Gasq D, De Boissezon X, Guillotreau J, Bourg V, Viala F, Rischmann P, Marque P. Urinary complications and risk factors in symptomatic multiple sclerosis patients. Study of a cohort of 328 patients. Neurourol Urodyn. 2015 Jan;34(1):32-6. doi: 10.1002/nau.22495. Epub 2013 Sep 23. PMID 24115110
- [Result] Castel-Lacanal E, Peyronnet B, Karsenty G, Loche CM, Phe V, Chartier-Kastler E, Cornu JN, Biardeau X, Even A, Denys P, Guinet-Lacoste A, Ruffion A, Bart S, Berard E, Game X. Evaluation of transcutaneous electrical tibial nerve stimulation in lower urinary tract dysfunction secondary to a parkinsonian syndrome: Uroparktens-a multicenter randomized placebo-controlled study. World J Urol. 2025 Apr 7;43(1):214. doi: 10.1007/s00345-025-05597-2. PMID 40192925